CLINICAL TRIAL: NCT05881343
Title: Retrospective Evaluation of Patients With Coronavirus 19 Infection Undergoing Major Orthopedic Urgent Surgery: a Case Series
Brief Title: Retrospective Case Series of COVID19+ Patients Undergoing Orthopedic Surgery
Acronym: COVID19&SURG
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: CORONAVIRUS&SURGERY
Record Dates: First submitted 2021-07-31; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2021-07

CONDITIONS: Coronavirus Infection; Orthopedic Disorder; Bone Fracture; Bone Metastases; Bone Neoplasm
Keywords: coronavirus; orthopedic surgery; SARS COV 2; COVID19
MeSH Terms: conditions — Coronavirus Infections; Musculoskeletal Diseases; Fractures, Bone; Bone Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Over the last months, the Rizzoli Orthopedic Institute in Bologna, Italy, has drained orthopedic urgencies from all other hospitals in the urban and suburban area. In this context urgencies are defined as fractures and primary or metastatic bone lesions with indication to non-deferrable surgery. A subset of these patients tested positive for SARS CoV 2, either before or after the surgical procedure.

Anesthesiological clinical management of covid19 cases is complicated by the consequences of the viral infection on respiratory and cardio-vascular systems, renal function and coagulation. Similarly, management of asymptomatic patients is challenging because of the lack of data on possible specific complications.

This study will report a snapshot of our early experience on perioperative clinical management of patients undergoing orthopedic surgery in the presence of SARS CoV 2 infection, ascertained or not at the time of surgery.

DETAILED DESCRIPTION:
This is a monocentric, retrospective, observational study.

the study will analyze all medical records of patients that underwent major or non-delayable orthopaedic surgery from the 1st of March 2020 to the 30th of June 2020 with known ongoing Coronavirus infection or postoperative diagnosis via nasal swab test collected at Rizzoli Orthopaedic Institute.

Medical history, anthropometrical, clinical, radiological, and biochemical data will be inserted in a database.

Primary objective will be to estimate population mortality in the time frame from surgery to hospital discharge.

Secondary objectives will be estimation of correlation between SARS-CoV2 infection and main postoperative complications. Mortality and site infection rate will be compared among the cohort and pre-COVID19 similar data.

Continuous variables will be summarized using median and interquartile range while dichotomic variables will be expressed as absolute and relative frequencies. Frequencies and outcomes will be reported as absolute frequency (observed / total) and relative percentage. Association between independent variables and outcomes will be tested with multivariate analysis, hypothesis testing (t-test or Mann-Whitney) and Fisher's exact test according to the type of variable and its distribution (and the experimental question at hand). Variables showing statistically significant association (p<0.1), will be used to build a multivariate logistic regression model with dichotomic dependent variable. Statistical significance threshold will be set to 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients urdergoing non-deferrable Orthopaedical surgery
* Ascertained SARS-CoV-2 infection detected by nasopharyngeal swab before of after the surgery
* Written, signed informed consent to the trial.

Exclusion Criteria:

* Lack of signed informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing non-deferrable Orthopaedic surgery (fractures, primary or metastatic bone lesions) in presence of SARS-CoV-2 infection, ascertained at the time of the surgery or detected by nasopharyngeal swab after the surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-07-18 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 infection | at baseline (day 0)
  Overall mortality in patients with ascertained SARS-CoV-2 infection undergoing major orthopaedic surgery
SARS-CoV-2 mortality | at baseline (day 0)
  Overall mortality in patients with ascertained SARS-CoV-2 infection undergoing major orthopaedic surgery

SECONDARY OUTCOMES:
Population | at baseline (day 0)
  Descriptive analysis of the characteristics of the population
Known SARS-CoV2 infection and type of anesthesia | at baseline (day 0)
  Correlation between known SARS-CoV2 infection at the time of surgery and type of anesthesia
Known SARS-CoV2 mortality | at baseline (day 0)
  Correlation between known SARS-CoV2 infection at the time of surgery and mortality
Known SARS-CoV2 infection | at baseline (day 0)
  Correlation between known SARS-CoV2 infection at the time of surgery and mortality
SARS-CoV2 infection and DVT/PE | at baseline (day 0)
  Correlation between ascertained SARS-CoV2 infection and deep vein thrombosis/pulmonary embolism
SARS-CoV2 and surgical site infection | at baseline (day 0)
  Correlation between ascertained SARS-CoV2 infection and surgical site infection
SARS-CoV2 and postoperative oxygen therapy | at baseline (day 0)
  Correlation between ascertained SARS-CoV2 infection and need for postoperative oxygen therapy / non-invasive or invasive ventilation
SARS-CoV2 infection and TEG | at baseline (day 0)
  Correlation between ascertained SARS-CoV2 infection and thromboelastography indicies.
Mortality in SARS-CoV2 patients vs historical population | at baseline (day 0)
  Comparison of mortality of patients with SARS-CoV2 infection with historical population data subjected to urgent orthopedic surgery.
Surgical site infection in SARS-CoV2 patients vs historical population | at baseline (day 0)
  Comparison of surgical site infection rate of patients with SARS-CoV2 infection with historical population data subjected to urgent orthopedic surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Bonarelli, MD, Principal Investigator — Post-operative Anaesthesia and Intensive Care and Pain Therapy - IRCCS Rizzoli Orthopaedic Institute
Locations (1):
- IORizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Publication or posting on trial registers

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Holshue ML, DeBolt C, Lindquist S, Lofy KH, Wiesman J, Bruce H, Spitters C, Ericson K, Wilkerson S, Tural A, Diaz G, Cohn A, Fox L, Patel A, Gerber SI, Kim L, Tong S, Lu X, Lindstrom S, Pallansch MA, Weldon WC, Biggs HM, Uyeki TM, Pillai SK; Washington State 2019-nCoV Case Investigation Team. First Case of 2019 Novel Coronavirus in the United States. N Engl J Med. 2020 Mar 5;382(10):929-936. doi: 10.1056/NEJMoa2001191. Epub 2020 Jan 31. PMID 32004427
- [Background] Silverstein WK, Stroud L, Cleghorn GE, Leis JA. First imported case of 2019 novel coronavirus in Canada, presenting as mild pneumonia. Lancet. 2020 Feb 29;395(10225):734. doi: 10.1016/S0140-6736(20)30370-6. Epub 2020 Feb 13. No abstract available. PMID 32061312
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Yu P, Zhu J, Zhang Z, Han Y. A Familial Cluster of Infection Associated With the 2019 Novel Coronavirus Indicating Possible Person-to-Person Transmission During the Incubation Period. J Infect Dis. 2020 May 11;221(11):1757-1761. doi: 10.1093/infdis/jiaa077. PMID 32067043
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Bai Y, Yao L, Wei T, Tian F, Jin DY, Chen L, Wang M. Presumed Asymptomatic Carrier Transmission of COVID-19. JAMA. 2020 Apr 14;323(14):1406-1407. doi: 10.1001/jama.2020.2565. PMID 32083643